CLINICAL TRIAL: NCT02781649
Title: An Open-label Pilot Study to Determine the Tolerability and Efficacy of Fixed-dose Grazoprevir/Elbasvir Treatment in Hepatitis C Uninfected Recipients of Renal Transplants From Hepatitis C Infected Deceased Donors
Brief Title: Exploring Renal Transplants Using Hepatitis C Infected Donors for HCV-negative Recipients
Acronym: EXPANDER-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00089751
Record Dates: First submitted 2016-05-10; First posted 2016-05-24 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: End-Stage Renal Disease; Hepatitis C
Keywords: Renal; Transplants; Hepatitis C; HCV-negative; Infected; Donors
MeSH Terms: conditions — Kidney Failure, Chronic; Hepatitis C | interventions — elbasvir-grazoprevir drug combination; grazoprevir; elbasvir; Ribavirin; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Donor genotype 1a no resistance or 1b (Experimental): Participants who receive donors found to have hepatitis C genotype 1a without resistance Zepatier one tablet daily for 12 weeks
  Interventions: Drug: Zepatier
- Donor genotype 1a with resistance (Experimental): Participants who receive donors found to have hepatitis C genotype 1a with nonstructural protein 5A associated resistance mutations Zepatier one tablet daily for 16 weeks Ribavirin weight based dosing for 16 weeks
  Interventions: Drug: Zepatier; Drug: Ribavirin
- Donor genotype 2 or 3 (Experimental): Participants who receive donors found to have hepatitis C genotype 2 or 3 Zepatier one tablet daily for 12 weeks Sofosbuvir 400 mg daily for 12 weeks
  Interventions: Drug: Zepatier; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Zepatier — Fixed dose Grazoprevir 100 mg/Elbasvir 50 mg by mouth daily for 12 weeks
  Other Names: Fixed dose Grazoprevir /Elbasvir
Drug: Ribavirin — Ribavirin 1200 mg/d (> 75 kg) or 1000 mg/d (< 75 kg) by mouth daily in two divided doses
  Other Names: Rebetol, Copegus, Virazole, and Ribasphere
  Arms: Donor genotype 1a with resistance
Drug: Sofosbuvir — Sofosbuvir 400 mg daily
  Other Names: Sovaldi
  Arms: Donor genotype 2 or 3

SUMMARY:
In this study, individuals without hepatitis C infection who are on the kidney transplant waitlist will receive a kidney from a deceased donor with hepatitis C infection and will be treated for hepatitis C at the same time. Treatment will include Grazoprevir (GZR) 100 mg/Elbasvir (EBR) 50 mg administered on-call to the operating room for the renal transplant procedure and continued for 12 weeks post-renal transplant.

DETAILED DESCRIPTION:
In this study, individuals without hepatitis C infection who are on the kidney transplant waitlist will receive a kidney from a deceased donor with hepatitis C infection and will be treated for hepatitis C at the same time. Hepatitis C treatment will include Grazoprevir (GZR) 100 mg/Elbasvir (EBR) 50 mg administered on-call to the operating room for the renal transplant procedure and continued for 12 weeks post-renal transplant. The donor hepatitis C genotype will be tested. If the donor has genotype 1a without resistance or genotype 1b treatment will remain GZR/EBR for 12 weeks. If the donor has genotype 1a with resistance variants, then Ribavirin will be added and treatment will be given for 16 weeks starting from the date ribavirin was added. If the donor has hepatitis C genotype 2 or 3, Sofosbuvir will be added and treatment will be for 12 weeks from the date Sofosbuvir was added.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 50 years old
* On the deceased donor kidney waiting list at Johns Hopkins Hospital
* Awaiting a first kidney transplant
* No available living kidney donors
* On hemodialysis or peritoneal dialysis or stage 5 chronic kidney disease (CKD) defined as a glomerular filtration rate < 15 ml/min for ≥ past 90 days
* HCV-uninfected (by both antibody and RNA PCR) and without any behavioral risk factors for contracting HCV other than being on hemodialysis.
* Calculated panel reactive anti-human leukocyte antigen (HLA) antibody (cPRA) below 20 percent
* Female who is:

  * practicing total abstinence from sexual intercourse (minimum 1 complete menstrual cycle)
  * sexually active with female partners only
  * not of childbearing potential: defined as postmenopausal for at least 2 years prior to screening defined as amenorrheic for longer than 2 years, age appropriate, and confirmed by a follicle-stimulating hormone level indicating a postmenopausal state, or surgically sterile: defined as bilateral tubal ligation, bilateral oophorectomy or hysterectomy or has a vasectomized partner(s);
  * of childbearing potential and sexually active with male partner(s): currently using at least one effective method of birth control at the time of screening and agree to practice two effective methods of birth control while receiving study drug (as outlined in the participant information and consent form starting with Study Day 1 and for 30 days after stopping study drug, or for 6 months after stopping study drug if receiving RBV (Note: Estrogen-containing hormonal contraceptives, including oral, injectable, implantable, patch and ring varieties, may not be used during study drug treatment).
* Males who are not surgically sterile and are sexually active with female partner(s) of childbearing potential must agree to practice two effective forms of birth control (as outlined in the participant information and consent form) throughout the course of the study, starting with starting with Study Day 1 and for 30 days after stopping study drug, or for 6 months after stopping study drug if receiving ribavirin (RBV)

Exclusion Criteria:

* Plan to receive a multi-organ transplant
* Plan to receive a dual kidney transplant (including en bloc)
* Prior solid organ transplant
* Participating in another study that involves an intervention or investigational product
* Plan to receive a blood type incompatible kidney
* History of human immunodeficiency (HIV), hepatitis C (HCV), or active hepatitis B (HBV) infection defined as being on active antiviral treatment for HBV, detectable hepatitis B surface Ag or detectable hepatitis B DNA
* Active or unresolved bacterial, viral, or fungal infection that is clinically significant
* History of cirrhosis or pre-existing liver disease such as non-alcoholic steatohepatitis
* History of illicit drug use or alcohol abuse within 12 months prior to screening
* Psychiatric or physical illness that in the opinion of the investigator would make it unsafe to proceed with transplantation or interfere with the ability of the subject to participate in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Peer reviewed publications

REFERENCES:
- [Derived] Durand CM, Bowring MG, Brown DM, Chattergoon MA, Massaccesi G, Bair N, Wesson R, Reyad A, Naqvi FF, Ostrander D, Sugarman J, Segev DL, Sulkowski M, Desai NM. Direct-Acting Antiviral Prophylaxis in Kidney Transplantation From Hepatitis C Virus-Infected Donors to Noninfected Recipients: An Open-Label Nonrandomized Trial. Ann Intern Med. 2018 Apr 17;168(8):533-540. doi: 10.7326/M17-2871. Epub 2018 Mar 6. PMID 29507971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
Started | 7 (4 in this group had insufficient viral RNA for genotyping. They were treated as 1a) | 0 | 3
Completed | 7 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were no participants who received a kidney from a donor with genotype 1a infection and resistance. Therefore this population is zero.
Groups:
- Total: Total of all reporting groups
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3 | Total
Number analyzed (Participants) | 7 | 0 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 2 | 2
  >=65 years | 7 | 0 | 1 | 8
Age, Continuous [Median (Full Range); unit: years] | 71 [65 to 76] |  | 61 [57 to 74] | 71 [57 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 6 | 0 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 6 | 0 | 2 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 |  | 3 | 10
Hepatitis C virus (HCV) antibody negative [Count of Participants; unit: Participants] | 7 | 0 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Higher Treatment-related Adverse Events as US Department of Health and Human Services Common Terminology of Adverse Events (CTCAE) Version 4
Description: Proportion of participants with grade 3 or higher treatment-related adverse events (AE) as assessed by US Department of Health and Human Services Common Terminology of AEs version 4. An AE is an unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5. Grade 3 Severe or medically significant but not life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE. The investigator will determine if the AE is related to the treatment.
Time Frame: 12 weeks after transplant
Population: There were no participants who received donors found to have hepatitis C genotype 1a with resistance enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
Number analyzed (Participants) | 7 | 0 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: Viral Response
Description: This is the number of participants with undetectable hepatitis C RNA in the blood at 12 weeks after stopping treatment. Proportion of kidney transplant recipients with HCV RNA < Lower Limit Of Quantification (LLOQ) at week 12
Time Frame: 12 weeks after completing treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
Number analyzed (Participants) | 7 | 0 | 3
Participants | 7 | 0 | 3

3. Secondary Outcome: Antibody Development
Description: Number of kidney transplant recipients who become reactive for HCV antibody
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
Number analyzed (Participants) | 7 | 0 | 3
Participants | 3 | 0 | 2

4. Secondary Outcome: Number of Participants With Nonstructural Protein 5A (NS5A) Resistance Mutations in the HCV Population From the Deceased Donors
Description: Number of participants with NS5A resistance mutations in the HCV population from the deceased donors.
  Number of donors with NS5A resistance mutations
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
Number analyzed (Participants) | 7 | 0 | 3
Participants | 0 | 0 | 0

5. Secondary Outcome: IP-10 Elevations
Description: Measurement of interferon (IFN)-gamma inducible protein 10 (IP-10) a marker of acute hepatitis C infection.
Time Frame: 12 weeks
Population: Data were not collected
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Kidney Function at 6 Months
Description: Serum creatinine mg/dL at 6 months following transplantation
Time Frame: 6 months following transplantation
Population: as for baseline characteristics
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
Number analyzed (Participants) | 7 | 0 | 3
mg/dL | 1.12 [1.06 to 1.7] |  | 0.9 [0.9 to 1.0]

7. Secondary Outcome: Kidney Function at 12 Months
Description: Serum creatinine mg/dL at 12 months following transplantation
Time Frame: 12 months following transplantation
Population: as for baseline characteristics
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
Number analyzed (Participants) | 7 | 0 | 3
mg/dL | 1.0 [0.9 to 1.0] |  | 1.3 [1.0 to 2.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 6 months from initiation of treatment
Description: 10 patients overall were at risk of adverse events, none of them from the Donor Genotype 1a With Resistance arm
Arm/Group | Donor Genotype 1a no Resistance or 1b | Donor Genotype 1a With Resistance | Donor Genotype 2 or 3
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/7 | 0/0 | 1/3
Other Adverse Events (participants affected / at risk) | 0/7 | 0/0 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor Genotype 1a no Resistance or 1b (N=7) | Donor Genotype 1a With Resistance (N=0) | Donor Genotype 2 or 3 (N=3)
Pulomonary infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
blood stream infection (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT02781649/Prot_SAP_001.pdf